CLINICAL TRIAL: NCT05193682
Title: Evaluation Of Right Ventricular Function In Septic Shock Patients In Intensive Care Unit.
Brief Title: Right Ventricular Dysfunction in Septic Shock Patients in ICU
Acronym: Septicshock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shimaa Hammad Ahmed (Other)
Responsible Party: Sponsor-Investigator, Shimaa Hammad Ahmed, Resident doctor at critical care unit, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Septic shock in ICU patients.
Record Dates: First submitted 2021-12-30; First posted 2022-01-18 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Assesment of right ventricular dysfunction in septic shock patients in intensive care unit.

DETAILED DESCRIPTION:
Over the last decade, a few studies have highlighted the crucial role of right ventricular (RV) function in hemodynamic and respiratory diseases in critical care 1,2. However, RV failure is difficult to define in the critical care setting. A recent consensual definition proposed by different groups of experts characterizes RV failure as the association of a significant RV dilatation associated with systemic congestion 3-5. This definition is mainly physiologically based, not strictly validated, and the experts did not propose any threshold for RV size or congestion using critical care echocardiography (CCE) and central venous pressure (CVP), respectively.

Fluid management in septic shock is crucial for prognosis, as fluid overload and high CVP are associated with a worse outcome 6. Septic shock is expected to impair RV function through the development of septic cardiomyopathy, but the incidence of RV failure is unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with septic shock.
2. Patients will be evaluated within 24 h after diagnosis.

Exclusion Criteria:

1. Patients diagnosed more than 24 hours.
2. Patients with associated ischemic heart failure .

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Septic shock patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Right ventricular dysfunction in septic shock patients in intensive care unit | 3 years
  Fluid management in septic shock is crucial for prognosis, as fluid overload and high CVP are associated with a worse outcome 6. Septic shock is expected to impair RV function through the development of septic cardiomyopathy, but the incidence of RV failure is unknown.